CLINICAL TRIAL: NCT02968836
Title: Safety and Efficacy of an Amino Acid Blend on Muscle and Gut Functionality in ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 15.04.CLI
Record Dates: First submitted 2016-10-19; First posted 2016-11-21 (Estimated); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Enteral Nutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Active Comparator): Blend of amino acids
  Interventions: Dietary Supplement: Blend of amino acids
- Placebo group (Placebo Comparator): maltodextrin only
  Interventions: Dietary Supplement: Maltodextrin only

INTERVENTIONS:
Dietary Supplement: Blend of amino acids — The product was poured in bottles containing the enteral nutrition that the patient received as standard of care.
  Arms: Active group
Dietary Supplement: Maltodextrin only — The product was poured in bottles containing the enteral nutrition that the patient received as standard of care.
  Arms: Placebo group

SUMMARY:
Assessment of the Safety and efficacy of an amino acid blend on muscle and gut functionality in Intensive Care Unit (ICU) patients.

Since this was a proof of concept, exploratory trial, we assessed different primary outcomes without hierarchy.

DETAILED DESCRIPTION:
This monocentric trial was a parallel, randomized, double-blind, controlled study. Patients hospitalized in the ICU for sepsis or ARDS were enrolled.

The treatment group (n=15) was administered the study product (amino acid blend) and the negative control group (=15) was administrated maltodextrin only. The mode of administration was nasogastric probe.

The treatment period was 21 days. Subject were followed during stay in High care and intermediate care units up to 2 months or after hospital discharge with a follow up until 12 months.

Recruitment stopped when 30 patients (15 in each group) reached V4.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 and over
2. Sepsis or ARDS patients: expected to stay at least 21 days in ICU (or midcare), to the opinion of the investigator
3. Informed consent signed by the patient or/and by his/her representative

Exclusion Criteria:

1. Patient with muscle mass loss due to previous hospitalization
2. Intolerance to enteral feeding
3. Patients using parenteral feeding
4. Chronic renal failure to the opinion of the investigator
5. Chronic liver disease to the opinion of the investigator
6. Cachectic patients
7. Current treatment with paralyzing drugs
8. No pacemaker or metal implants interacting with MRI and magnetic stimulation
9. Pregnant woman (known)
10. Persons without social security
11. Under guardianship
12. Currently participating or having participated in another clinical trial within 4 weeks prior to trial start
13. Patient who is expected not to comply with the study procedures, to the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Safety: Renal function change | 60 days from the beginning of the intervention
  Renal function will be daily assessed from urine output, serum creatinin and glomerular filtration rate
Efficacy: muscle functionality change | 12 months from the beginning of the intervention (timepoints: D1, D7, D14, D21, D60, D180, D365)
  i. Muscle (quadriceps) extension isometric strength in response to magnetic stimulation; diaphragm muscle strength in response to magnetic stimulation. Forced vital capacity and maximal inspiratory and expiratory pressures will systematically be recorded.
  ii. Loss in quadriceps muscle mass and metabolism will be measured by Magnetic resonance imaging.
  Muscle protein catabolism will be evaluated from measures of 3-methyl histidine in the 24-h urine (reported to urine creatinine).
Efficacy: gut barrier structure and functionality improvement | 12 months from the beginning of the intervention (timepoints: D1, D7, D14, D21, D60, D180, D365)
  i. Enterocytes damage by measurement of I-FABP (intestinal fatty acid-binding protein) in plasma and urine.
  ii. Functional enterocyte mass by citrulline plasma concentration. iii. Gut barrier function by the translocation of bacteria based on plasma D-Lactate concentration
Efficacy: inflammatory status change | 12 months from the beginning of the intervention (timepoints: D1, D7, D14, D21, D60, D180, D365)
  i. Calprotectin in feces, which is secreted by the neutrophils of the gut mucosae and is released in the gut when the mucosa is inflamed.
  ii. Acute phase protein concentration in plasma (CRP, fibrinogen, ferritin, prealbumin)
Efficacy: general recovery improvement | 12 months from the beginning of the intervention (timepoints: D1, D7, D14, D21, D60, D180, D365)
  i. Length of stay (LOS) in High care and intermediate care units. ii. Time (days) free of ventilation until discharge high care. iii. Time (days) to recover on walking with or without aid
Nutrient profiling | Over 60 days from the beginning of intervention (timepoints: D1, D7, D14, D21, D60)
  Nutrient profiling will be assessed from blood metabolomics analyses

CONTACTS AND LOCATIONS:
Overall Officials: Djillali Annane, Pr, Principal Investigator — Raymond Poincaré Hospital, Garches, France
Locations (1):
- Hôpital Raymond Poincaré (AP-HP), Garches, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heming N, Carlier R, Prigent H, Mekki A, Jousset C, Lofaso F, Ambrosi X, Bounab R, Maxime V, Mansart A, Crenn P, Moine P, Foltzer F, Cuenoud B, Konz T, Corthesy J, Beaumont M, Hartweg M, Roessle C, Preiser JC, Breuille D, Annane D. Effect of an enteral amino acid blend on muscle and gut functionality in critically ill patients: a proof-of-concept randomized controlled trial. Crit Care. 2022 Nov 17;26(1):358. doi: 10.1186/s13054-022-04232-5. PMID 36397118